CLINICAL TRIAL: NCT02892188
Title: Assessment of the Follow-up of Osteoporotic Patients by a Physician-pharmacist Collaboration
Brief Title: Physician-Pharmacist Collaboration for Osteoporotic Patient Follow-up
Acronym: SIOUX
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-01Obs-CHRMT
Record Dates: First submitted 2016-08-26; First posted 2016-09-08 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the follow-up of the osteoporotic patient by a physician-pharmacist collaboration.

DETAILED DESCRIPTION:
Treatments allow decreasing the personal fracture risk from 48% to 85% provided that the treatment period is continued at least 3 to 5 years and that hygienic and dietary measures are applied: optimization of the dietary calcium intakes (much more efficient and less dangerous than the medicinal intakes), preservation of a physical activity, fall prevention. The ability of bisphosphonate for decreasing significantly the number of fractures was proved, but the lack of lasting adhesion (persistence) and of flanking measures leads to believe their efficiency may be enhanced: the hip-fracture rate decreases from 2.1% for the non-adherents to 1,3% for the patients with observance, which represents a one-half reduction.

The cost of surgery for a femoral neck fracture is estimated at 8500 euros. So the prevention of only one femoral neck fracture entails a huge economy.

However, 50% of women stop their treatment before a year and the implementation of hygienic and dietary measures leads to a lifestyle change, and faces long time ingrained habits. Only 42% of patients continue their treatment after two years, and only 16% after three years.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years old
* having an osteoporosis treatment
* following a Therapeutical Education for Patient

Exclusion Criteria:

* opposition for anonymised data gathering

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient having osteoporosis enrolled into the programm of Therapeutical Educational for patient
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Respect of treatment and of hygienic dietary measures by patients with a self-questionnaire per medical check | year 3
  This assessment will be made at the end of the follow-up, after three years, but an intermediary assessment about those same criteria is planned at one and two years of the follow-up.

SECONDARY OUTCOMES:
Qualitative evaluation of the professional adhesion for the follow-up process once a year during the annual meeting | year 3
  This assessment will be made at the end of the follow-up, after three years, but an intermediary assessment about those same criteria is planned at one and two years of the follow-up.
Quantitative evaluation of it by the return rate of questionnaires | year 3
  This assessment will be made at the end of the follow-up, after three years, but an intermediary assessment about those same criteria is planned at one and two years of the follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Didier POIVRET, MD, Principal Investigator — CHR Metz-Thionville
Locations (1):
- CHR Metz-Thionville, Metz, France

IPD SHARING:
Plan to Share IPD: No